CLINICAL TRIAL: NCT00342849
Title: Treatment of Lead-Exposed Children (TLC) Trial
Brief Title: Treatment of Lead-Exposed Children Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 999994037; OH94-E-N037
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2015-06-10

CONDITIONS: Lead Exposure
Keywords: Clinical Trial; Low-level Lead Poisoning; Chelation; Developmental Assessment; Succimer
MeSH Terms: interventions — Succimer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Experimental): Scuccimer Treatment Group
  Interventions: Drug: Succimer
- 2 (Placebo Comparator): In order to provide placebo with an odor comparable to that of succimer, the Drug Distribution Center will place a small canister containing 200 mg of active drug into each bottle of placebo drug. A canister containing 200 mg of placebo will be placed inside each bottle of succimer so that all bottles will appear the same.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Succimer — Succimer (2,3-meso-dimercaptosuccinic acid) is an orally active dithiol compound that is a relatively specific chelating agent for heavy metals, especially lead, arsenic and mercury. The drug undergoes limited absorption in the gastrointestinal tract and then is rapidly metabolized to mixed disulfides which are eliminated in the urine. Blood levels decline slowly with an apparent elimination half-life of about 48 hours in adults.
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The Treatment of Lead-Exposed Children (TLC) clinical trial compared the effect of lead chelation with succimer to placebo therapy. TLC was a randomized, double-blind, placebo-controlled clinical trial with sites in Cincinnati and Columbus, Ohio, Philadelphia, Pennsylvania, Baltimore, Maryland and Newark, New Jersey. The study was designed to test outcomes in IQ, neuropsychological function, behavior, physical growth and blood pressure three years after initiation of treatment. Enrollment was conducted between 1994 and 1997, with completion of the initial three-year follow-up in 2000.

DETAILED DESCRIPTION:
At TLC enrollment, the children were between 12 and 33 months of age with baseline blood lead levels (PbB) between 20 and 44 microg/dl. Of 1,854 referred children who were screened for eligibility, 780 were randomized to the active drug (oral succimer) and placebo groups, stratified by clinical center, body surface area, blood lead level and language spoken at home; only the New Jersey Clinical Center enrolled Spanish-speaking participants. Up to three 26-day courses of succimer or placebo therapy were administered depending on response to treatment in those who were given the active drug. Eighty-nine percent of children had finished treatment by six months, with all children finishing by 13 months after randomization. Residential lead clean-up and nutritional supplementation with multivitamins and minerals were provided to all study children, irrespective of treatment group. Children were followed for three years, with regular physical exams, psychological and developmental testing, and measurement of lead concentration in venous blood. Treatment and follow up are closed for this trial; it is open for scientific analysis and report writing only.

Although succimer lowered blood lead levels much more effectively than placebo, there was no difference between the two groups on any of the psychological tests at three years post randomization, when most children were about five years old. Follow up of TLC children continued into school age. At age seven, 647 of 780 subjects remained in the study. Children were tested at age seven and again at seven and a half on standardized neuropsychological batteries that tap cognition, behavior, learning and memory, attention, and neuromotor skills. While chelation therapy with succimer had lowered average blood lead levels for approximately six months, it resulted in no benefit in cognitive, behavioral and neuromotor endpoints when measured at school ages in these children. These additional follow-up data confirm our previous finding that the TLC regimen of chelation therapy is not associated with neurodevelopmental benefits in children with blood lead levels between 20 and 44 microg/dL.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study population will reflect the population known to be at greatest risk to lead exposure, i.e., low income, urban, African-American children.

EXCLUSION CRITERIA:

Linguistic minorities will be excluded in all centers except Newark, where Hispanic children make up a sizable portion of the population and will be included.

Ages: 12 Months to 33 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 780 (Actual)
Dates: Start 1994-07-15; Primary Completion 2007-08-29 (Actual); Study Completion 2015-06-10 (Actual)

PRIMARY OUTCOMES:
Efficacy | Annually

CONTACTS AND LOCATIONS:
Overall Officials: Walter Rogan, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (4):
- United States (4):
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Childrens Hospital, Columbus, Columbus, Ohio
  - Childrens Hospital, Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Littman E, Goldstein MH, Kasen L, Levitt MF, Wedeen RP. The relationship of the intrarenal distribution of Hg203-chlormerodrin to the diuretic effect. J Pharmacol Exp Ther. 1966 Apr;152(1):130-8. No abstract available. PMID 5937397
- [Background] Levitt MF, Goldstein MH, Lenz PR, Wedeen R. Mercurial diuretics. Ann N Y Acad Sci. 1966 Nov 22;139(2):375-87. doi: 10.1111/j.1749-6632.1966.tb41211.x. No abstract available. PMID 5230281
- [Background] Wedeen RP, Jernow HI. Autoradiographic study of cellular transport of hippuran-125I in the rat nephron. Am J Physiol. 1968 Apr;214(4):776-85. doi: 10.1152/ajplegacy.1968.214.4.776. No abstract available. PMID 5642938
- [Derived] Cao Y, Chen A, Bottai M, Caldwell KL, Rogan WJ. The impact of succimer chelation on blood cadmium in children with background exposures: a randomized trial. J Pediatr. 2013 Aug;163(2):598-600. doi: 10.1016/j.jpeds.2013.03.009. Epub 2013 Apr 16. PMID 23601497
- [Derived] Cao Y, Chen A, Jones RL, Radcliffe J, Dietrich KN, Caldwell KL, Peddada S, Rogan WJ. Efficacy of succimer chelation of mercury at background exposures in toddlers: a randomized trial. J Pediatr. 2011 Mar;158(3):480-485.e1. doi: 10.1016/j.jpeds.2010.08.036. PMID 20889164